CLINICAL TRIAL: NCT01066195
Title: A Phase III, Multi-center, Randomized Trial of Pemetrexed and Gefitinib in Never-smoker and Adenocarcinoma Patients With Non-small Cell Lung Cancer Previously Treated With Platinum-based Chemotherapy
Brief Title: Pemetrexed (ALIMTA) and Gefitinib (IRESSA®) in Never-Smoker and Adenocarcinoma Patients With Non-Small Cell Lung Cancer Previously Treated With Platinum-Based Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Samsung Medical Center (Other)
Responsible Party: Myungju Ahn Ph.D., M.D., Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-04-030
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2010-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Non-Small Cell Lung Cancer; Never-Smoker and Adenocarcinoma patients; Pemetrexed (ALIMTA); Gefitinib (IRESSA®)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib; Pemetrexed

ARMS (2):
- gefitinib (Experimental)
  Interventions: Drug: iressa
- pemetrexed (Active Comparator)
  Interventions: Drug: alimta

INTERVENTIONS:
Drug: iressa — iressa 250mg per day every day
  Arms: gefitinib
Drug: alimta — alimta 500mg/m2 every 3 weeks
  Arms: pemetrexed

SUMMARY:
Pemetrexed was known to be effective to pulmonary adenocarcinoma and gefitinib was known to be more effective to non-small cell lung cancer (NSCLC) patients with clinical characteristics such as adenocarcinoma, never smoker and female.

The investigators try to evaluate which drug (pemetrexed vs gefitinib) is more efficious to NSCLC patients with clinical characteristics such as adenocarcinoma and never smoking history as second- or further-line therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed pulmonary adenocarcinoma including bronchioloalveolar, but except adenosquamous cell carcinoma
2. Stage IIIB (malignant pleural effusion and/or pleural seeding), stage IV and relapsed non-small cell lung cancer
3. Failed with 1st line platinum-based chemotherapy or relapsed within 12 months after adjuvant platinum-based chemotherapy)
4. Never smoker (less than 100 cigarette for the life time)
5. 18 year or older
6. ECOG 0-2
7. No history of biologic or immunotherapy
8. Tolerable renal function ( creatine clearance rate is 60ml/min or more)
9. Tolerable hepatic function (Serum bilirubin ≤ 1.25 x UNL, AST (SGOT) and ALT (SGPT) ≤ 2.5 x UNL, alkaline phosphatase ≤5 x UNL)

Exclusion Criteria:

1. symptomatic brain metastasis
2. previously treated with EGFR tyrosine kinase inhibitor
3. previously treated with antifolate agents
4. poor oral absorption
5. patients with active infection
6. uncontrolled diabetes mellitus
7. significant cardiovascular disease (uncontrolled hypertension, history of myocardial infarction or unstable angina within 6 months, congestive heart failure)
8. pregnant or nursing patients
9. history of malignant disease within 3 years before the enrollment except for cured non-melanomatous skin cancer, cervical carcinoma in situ, or thyroid carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 36 months

SECONDARY OUTCOMES:
overall survival | 36 months
objective response rate | 36 months
toxicity | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Myungju Ahn, Ph.D., M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea